CLINICAL TRIAL: NCT05572099
Title: ExoDx Prostate Evaluation in Active Surveillance Patient Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Exosome Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECT2022-01
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ExoDx Prostate — Observational only.

SUMMARY:
The goal of this observational study is to test whether the ExoDx Prostate test add value in biopsy decision making to patients with prostate cancer on an active surveillance regimen.

DETAILED DESCRIPTION:
The current trial seeks to evaluate the role of the ExoDx Prostate test in men with low and favorable intermediate prostate cancer undergoing an active surveillance regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male, 45+ years of age diagnosed with low-grade or favorable-intermediate prostate cancer and on an active surveillance regimen

Exclusion Criteria:

* Clinical symptoms of urinary tract infection at time of enrollment.
* History of invasive treatment for benign prostatic hypertrophy with in 6 months of enrollment.
* Known hepatitis or HIV
* History of concurrent renal/bladder tumors

Min Age: 45 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Have a prostate
Study Population: Male, 45+ years of age diagnosed with low-grade or favorable-intermediate prostate cancer and on an active surveillance regimen
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Develop and evaluate risk-based scoring using the ExoDx Prostate test. | 1yr after last enrolled patient

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Kumar, PhD, Study Director — Exosome Diagnostics, Inc.
Locations (1):
- Chesapeake Urology, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided